CLINICAL TRIAL: NCT02555332
Title: Maternal TSH Level and TPOAb Status in Early Pregnancy and Their Relationship to the Risk of Gestational Diabetes Mellitus
Brief Title: Maternal Thyroid Function in Early Pregnancy and Their Relationship With Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Hao Ying, Director,Clinical research, Shanghai First Maternity and Infant Hospital
Other Study IDs: REB#12-054
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy; Thyroid Function Tests; Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women underwent screening for thyroid function: All these women underwent screening for thyroid function (TSH,FT4,TPOAb) at the first antenatal visit and the 75g oral glucose tolerance test (OGTT) at 24-28 weeks of gestation. The correlation between the combination of TSH level and TPOAb status and the risk of Gestational Diabetes Mellitus was analyzed.
  Interventions: Other: 75g oral glucose tolerance test (OGTT)

INTERVENTIONS:
Other: 75g oral glucose tolerance test (OGTT) — All these women underwent the 75g oral glucose tolerance test (OGTT) at 24-28 weeks of gestation.

SUMMARY:
This study was conducted to analyze the role of TSH level and TPOAb status in early pregnancy and use this information in assessment of the risk of gestational diabetes mellitus at different weeks of gestation when the FT4 level is normal.

DETAILED DESCRIPTION:
A total of 7,729 women with singleton pregnancies who were receiving antenatal care at Shanghai First Maternity and Infant Hospital, Tongji University School of Medicine between December 2012 and March 2014 were included in the study. All these women underwent screening for thyroid function (TSH,FT4 and TPOAb) at the first antenatal visit and a 75 g oral glucose tolerance test at 24-28 weeks of gestation. The correlation between a combination of TSH level and TPOAb status and the risk of gestational diabetes mellitus was analyzed.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

1. ≤19+6 weeks of gestation at the first antenatal visit;
2. singleton pregnancy;
3. FT4 level is within the normal range;
4. TSH level is normal or beyond the normal range.

Exclusion Criteria:

1. age <18 years or >40 years;
2. thyroid disease history before pregnancy, e.g. hyperthyroidism, clinical hypothyroidism and malignant tumors of the thyroid, regardless of medication treatment is needed or not;
3. twin or multiple gestations;
4. diagnosed with diabetes mellitus before pregnancy, or fasting blood-glucose level ≥ 7.0 mmol/L or HbA1C≥6.5% at the first antenatal visit;
5. diseases causing abnormal glycometabolism or severe co-morbidities or diseases causing abnormal glycometabolism.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the pregnant women who were receiving antenatal care at Shanghai First Maternity and Infant Hospital, Tongji University School of Medicine were invited to participate in the study.Informed consents were obtained from all subjects.
Sampling Method: Probability Sample
Enrollment: 7729 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
75g oral glucose tolerance test (OGTT) positive or not | 24-28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hao Ying, PHD, Principal Investigator — Shanghai First Maternity and Infant Hospital

REFERENCES:
- [Result] Agarwal MM, Dhatt GS, Punnose J, Bishawi B, Zayed R. Thyroid function abnormalities and antithyroid antibody prevalence in pregnant women at high risk for gestational diabetes mellitus. Gynecol Endocrinol. 2006 May;22(5):261-6. doi: 10.1080/09513590600630470. PMID 16785147
- [Result] Pascual Corrales E, Andrada P, Auba M, Ruiz Zambrana A, Guillen Grima F, Salvador J, Escalada J, Galofre JC. Is autoimmune thyroid dysfunction a risk factor for gestational diabetes? Endocrinol Nutr. 2014 Aug-Sep;61(7):377-81. doi: 10.1016/j.endonu.2014.01.009. Epub 2014 Mar 26. English, Spanish. PMID 24680382
- [Result] Tudela CM, Casey BM, McIntire DD, Cunningham FG. Relationship of subclinical thyroid disease to the incidence of gestational diabetes. Obstet Gynecol. 2012 May;119(5):983-8. doi: 10.1097/AOG.0b013e318250aeeb. PMID 22525909
- [Result] Olivieri A, Valensise H, Magnani F, Medda E, De Angelis S, D'Archivio M, Sorcini M, Carta S, Baccarini S, Romanini C. High frequency of antithyroid autoantibodies in pregnant women at increased risk of gestational diabetes mellitus. Eur J Endocrinol. 2000 Dec;143(6):741-7. doi: 10.1530/eje.0.1430741. PMID 11124856
- [Result] Karakosta P, Alegakis D, Georgiou V, Roumeliotaki T, Fthenou E, Vassilaki M, Boumpas D, Castanas E, Kogevinas M, Chatzi L. Thyroid dysfunction and autoantibodies in early pregnancy are associated with increased risk of gestational diabetes and adverse birth outcomes. J Clin Endocrinol Metab. 2012 Dec;97(12):4464-72. doi: 10.1210/jc.2012-2540. Epub 2012 Sep 26. PMID 23015651